CLINICAL TRIAL: NCT06633289
Title: Hypoallergenicity of a Hydrolyzed Rice Protein-based Formula in Infants and Young Children With Cow's Milk Protein Allergy: a Randomized Nutritional Clinical Study
Brief Title: Hypoallergenicity of a Hydrolyzed Rice Protein-based Formula in Infants and Young Children With Cow's Milk Protein Allergy
Acronym: RIGHT-HY
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: 2115INF
Record Dates: First submitted 2024-10-07; First posted 2024-10-09 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Cow's Milk Protein Allergy
MeSH Terms: conditions — Milk Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental formula-Control formula (Other): Blinded cross-over oral food challenge sequence starting by Experimental formula followed by Control.
  Following the crossover phase, children who passed the oral food challenge will consume the open label experimental formula at home during 7 days.
  Interventions: Other: Experimental formula; Other: Control formula
- Control formula-Experimental formula (Other): Blinded cross-over oral food challenge sequence starting by Control followed by Experimental formula.
  Following the crossover phase, children who passed the oral food challenge will consume the open label experimental formula at home during 7 days.
  Interventions: Other: Experimental formula; Other: Control formula

INTERVENTIONS:
Other: Experimental formula — New hydrolyzed rice protein-based formula
Other: Control formula — Commercially available amino acid-based formula.

SUMMARY:
The purpose of the study is to determine whether a new hydrolyzed rice protein-based formula is hypoallergenic in infants and young children with documented Immunoglobulin E (IgE)-mediated Cow Milk Protein Allergy (CMPA).

ELIGIBILITY:
Inclusion criteria:

1. Written informed consent has been obtained from at least one parent (or legally acceptable representative [LAR]), if applicable)
2. Child gestational age ≥ 37 completed weeks
3. Child aged ≥ 60 days and less than 36 months at enrollment
4. Documented IgE-mediated CMPA no more than 6 months prior to enrollment
5. Child is receiving a strict cow's milk elimination diet and will continue receiving this diet until the completion of the study
6. Child's parent(s) and LAR (if applicable) is of legal age of majority, must have parental authority, must understand the informed consent form and other study documents, and are willing and able to fulfill the requirements of the study protocol

Exclusion criteria:

1. Child is exclusively breastfed
2. Any chronic medical diseases (except atopic eczema), chromosomal or major congenital anomalies
3. Congenital heart disease or treatment by B-blockers
4. Major gastrointestinal disease / abnormalities (other than CMPA)
5. Known or suspected soy allergy
6. Glucose-galactose malabsorption
7. Immunodeficiency
8. Children who are unable to discontinue antihistamine use (excluding eye drops) within 7 days prior to a food challenge and oral steroid use within 14 days prior to enrollment
9. Persistent wheeze or chronic respiratory disease
10. Severe uncontrolled eczema or urticaria
11. Rice protein allergy or intolerance (e.g., rice protein-induced enterocolitis syndrome), or allergy to any ingredient in the formulas
12. Child's parent has other medical or psychiatric condition that, in the judgement of the Investigator, would make the child inappropriate for entry into the study
13. Currently participating or having participated in another interventional clinical study within 4 weeks prior to enrollment
14. Child's parents have not reached legal age of majority (18 years).

Ages: 60 Days to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Hypoallergenicity of a Hydrolyzed Rice Protein-based Formula (Experimental Formula) | during test day
  by measuring the proportion of participants who "passed" the food challenge test, meaning who consumed all doses and exhibited no allergic reactions to any of the doses of the experimental formula.

SECONDARY OUTCOMES:
Gastrointestinal tolerance of experimental formula during at home consumption period | during 7 days
  by evaluating gastrointestinal symptoms, using information recorded by parents daily in a diary
Safety of experimental formula during the at-home consumption | during 7 days
  By assessing the frequency and severity of adverse events reported by parents during the home usage phase

CONTACTS AND LOCATIONS:
Locations (11):
- Charité - Universitätsmedizin Berlin Klinik für Pädiatrie m.S. Pneumologie/Immunologie, Berlin, Germany
- Italy (4):
  - IRCCS Azienda Ospedaliero Universitaria Meyer Viale Gaetano Pieraccini, Florence
  - Ospedale dei Bambini V. Buzzi Via Castelvetro, 32, Milan
  - Universiy of Naples Federico II, Naples
  - Azienda Ospedaliero Universitaria di Parma, Italy, Parma
- Poland (6):
  - Nicolaus Copernicus University in Torun, Bydgoszcz
  - Centrum Medyczne Plejady, Krakow
  - Jagiellonian University Medical College, Krakow
  - Wojewodzki Szpital Specjalistyczny im. M. Kopernika, Lodz
  - BioMedical Centers sp. z o.o., Warsaw
  - Pediatrics Department at the Medical University of Warsaw, Warsaw

IPD SHARING:
Plan to Share IPD: No